CLINICAL TRIAL: NCT05936528
Title: The Effect of Lactoferrin in Improving Clinical Outcomes in ICU Patients
Brief Title: Lactoferrin Use in ICU Patients
Acronym: RCT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed H Hassan, PharmD, Principal Investigator, King Salman International university
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MD.23.09.800; 35039/9/23 (Other: Tanta University)
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Critical Illness
Keywords: Clinical outcomes; ICU patients; Lactoferrin; Antioxidant therapy; Anti-inflammatory therapy; Antimicrobial therapy
MeSH Terms: conditions — Critical Illness | interventions — Lactoferrin; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactoferrin (Experimental): Lactoferrin 100 mg sachets with a dose of 200 mg (2 sachets) orally twice daily (400 mg per day) In addition to standard of care
  Interventions: Drug: Lactoferrin
- Standard (Active Comparator): Subgroup B1 will receive standard antioxidant drug (Acetyl cysteine 600 mg / 12 hr) orally to be compared with lactoferrin A1 subgroup.
  * Subgroup B2 will receive standard anti-inflammatory, and immunomodulatory drug (dexamethasone I.V 8 mg / day) to be compared with lactoferrin A2 subgroup.
  * Subgroup B3 will receive standard antibacterial drugs to be compared with lactoferrin A3 subgroup.
  Interventions: Drug: Antioxidant therapies; Drug: Dexamethasone; Drug: Antibacterial therapies

INTERVENTIONS:
Drug: Lactoferrin — antioxidant, immunomodulatory, anti-inflammatory, antimicrobial effect
  Arms: Lactoferrin
Drug: Antioxidant therapies — Acetyl cysteine 600 mg / 12 hr
  Arms: Standard
Drug: Dexamethasone — dexamethasone I.V 8 mg / day
  Arms: Standard
Drug: Antibacterial therapies — Antibacterial drugs in their approved doses
  Arms: Standard

SUMMARY:
Introduction:

Lactoferrin has several uses due to its effects. It has anti-inflammatory, antioxidant, immunomodulatory, antibacterial, antifungal, and antiviral effects. Its safety is proven by food and drug administration.

Aims:

The objective is to study the effect of lactoferrin on improving clinical outcomes in ICU patients, and also to evaluate its safety.

Patients and populations:

A sample of 660 patients (330 patients in both groups A, and B) who will be admitted to ICU departments in Mansoura university hospital will be used to represent the population in ICU.

Methods:

A sample of 660 participants was randomized 1:1 into two groups (group A (330 patients), and group B (330 patients)).

This study is a single blind, randomized controlled clinical trial. Randomization was performed by independent clinical pharmacists working in hospital ICU departments.

DETAILED DESCRIPTION:
1. Introduction

   1.1. Lactoferrin molecule

   Lactoferrin (LF) is iron linking milk protein. LF helps to modulate iron levels in the body [1-3]. LF is a part of the milk whey protein. The colostrum (the first milk produced by mothers after delivery) has seven times more LF than mature milk [4]. LF is found in many organs like kidneys, lungs, gallbladder, pancreas, intestine, liver, prostate, and also in the body fluids like saliva, tears, sperm, cerebrospinal fluid, urine, bronchial secretions, vaginal discharge, synovial fluid, umbilical cord blood, blood plasma, and immune cells [1,2,4]. LF has many beneficial effects in the body. It has antioxidant, immunomodulatory, anti-inflammatory, antimicrobial, and antiviral effects [5]. Figure 1: different effects of lactoferrin [5]

   1.2. Lactoferrin as antioxidant molecule

   The body is affected by several factors such as pathogens, environmental pollutants, and toxins. This leads to the development and accumulation of reactive oxygen species (ROS) in the body which is known as oxidative stress. ROS can cause many diseases. LF can stop the harm induced by ROS [6, 7], and enhance the activity of endogenous antioxidant pathways [8].

   LF acts as a neuroprotective agent in Parkinson's disease and Alzheimer's disease [9]. It also protects against osteoporosis by inhibition of osteoblast activity and due to its antioxidant effect [10]. LF improves glucose metabolism in patients with type 2 diabetes mellitus via enhancement of the insulin-mediating response [11] and prevents obesity due to imbalance in body fat metabolism [12]. It also reduces blood pressure in hypertension [13]. So, LF can act as anti-hyperglycemic, and anti-hypertensive agent.

   1.3. Lactoferrin as antipathogenic and immunomodulating molecule LF has antibacterial activity against Gram-positive and Gram-negative bacteria, as it kills pathogens, and prevents the biofilm formation by Staphylococcus aureus or Pseudomonas aeruginosa [14]. LF also prevents viral, bacterial, fungal and protozoal gastrointestinal tract infections [15]. It enhances the treatment of Helicobacter pylori gastric infection [16], and also protects against endotoxemia, bacteremia, sepsis and necrotic enteritis after partial bowel resection [17] and in neonates [18]. LF possess an antiviral activity and enhances the effect of antiviral drugs [19].

   It acts as antiviral agent by blocking the pathogen's surface receptors and prevents it from binding to the target cell, for example, its binding to angiotensin converting enzyme II receptors which used by SARS-CoV-2 to pass cell membrane and thus inhibit virus entry into the cell [20].

   LF also has antifungal effect against dermatophytes and enhance the effect of antifungal drugs [21]. In addition, it has an antiparasitic effect in treatment of toxoplasmosis and malaria [22].

   It also has an immunomodulating effect, stimulating the body to synthesize cytokines and chemokines as well as accelerating the maturation of the immune system cells [3, 23].

   LF possesses also anti-inflammatory activity in non-infectious disorders such as allergies, arthritis, cancer [24] and inflammatory colitis [25]. Its anti-inflammatory effect is due to the inhibition of ROS to prevent lipid peroxidation by chelating iron. It also enhances the production of anti-inflammatory cytokines (IL-10) and suppresses the production of pro-inflammatory cytokines (IL-6, IL-8, IL-1b, and TNF-α). In addition, It can enter into mast cells and interact with the inflammatory proteases (chymase, cathepsin G, and tryptase) [26].

   1.5. Lactoferrin for anemia of inflammation

   LF treats inflammatory disorders by increasing ferroprotein production and decreasing IL-6 level to redistribute endogenous iron between blood and tissue. So, LF is used as therapy for anemia caused by inflammation [27].

   1.6. Safety of lactoferrin use

   The safety of LF is proved by the Food and Drug Administration. However, bovine LF, as an ingredient in cow's milk, may cause hypersensitivity, So, lactoferrin use has a risk of allergic reaction, and contraindicated in case of hypersensitivity to cow's milk proteins, and in lactose intolerance [28]. Other side effects of LF include stomach pain, vomiting, and constipation [29].
2. Aim of the study

   The objective is to study the effect of lactoferrin on improving clinical outcomes in ICU patients, and also to evaluate its safety.
3. Methods

   3.1. Study design

   The research will be a single-blind, randomized, controlled clinical trial to evaluate the efficacy and safety of a drug. Randomization will be 1:1 and achieved by independent clinical pharmacists who are working in ICU departments of the hospital. The patients will be blinded for identification of treatment, and placebo groups. Allocation of patients into their groups will be made after checking for meeting inclusion and not meeting exclusion criteria within 24 hours of the admission to ICU. All patients will receive the standard of care at admission.

   3.2. Patients and populations

   A total of 660 patients who will be admitted to ICU departments in Mansoura University Hospital will represent the population in ICU.

   3.3. Intervention

   One group will receive a two sachet of 100 mg lactoferrin enterally (either orally or by Ryle tube) every 12 hours (400 mg daily) for 28 days plus the standard of care. another group will receive the standard of care only.

   A sample of 660 patients (330 patients in both 2 groups (group A: lactoferrin and group B: standard group) who will be admitted to ICU departments in Mansoura university hospital will be used to represent the population in ICU. The standard group (B) will be divided into three subgroups of 110 patients in each. Subgroup B1 will receive standard antioxidant drug (Acetyl cysteine 600 mg / 12 hr) orally to be compared with lactoferrin A1 subgroup.

   - Subgroup B2 will receive standard anti-inflammatory, and immunomodulatory drug (dexamethasone I.V 8 mg / day) to be compared with lactoferrin A2 subgroup.
   * Subgroup B3 will receive standard antibacterial drugs to be compared with lactoferrin A3 subgroup.

   3.4. Outcomes and parameters

   Primary outcomes:
   * 28-day mortality (efficacy), and
   * incidence of any allergic or hypersensitivity reactions (safety).

   Secondary outcomes:

   • the day of death,

   • need for invasive mechanical ventilation (IMV),

   • duration of need for oxygen therapy, and IMV,

   • duration of ICU stay, and

   • kidneys, and liver functions.

   • Glasgow coma score (GCS) and

   • sequential organ function assessment (SOFA) score [31].

   • The changes in biochemical markers

   Blood sample collection:

   About 5 ml venous blood samples will be withdrawn by sterile venipuncture and centrifugated at 3000 rpm for 15 min, then sera will be kept frozen at 8 oC until analysis of • CBC • Inflammatory marker (TNF-α) • Oxidant marker (TAC)
   * Liver functions
   * Kidney functions In addition, arterial blood gases (ABG), vital signs, and Oxygen saturation were measured.Most of these parameters are measured in previous researches [32-39]

   Subgroup analysis will be conducted in order to compare lactoferrin with other drugs with relevant activity as shown below:

1- A comparison between the adjuvant antibacterial effect of lactoferrin vs standard antibacterial drugs as indicated by the WBCs and its differential counts (neutrophils, macrophages) in case of bacterial infections.

2- A comparison between the antioxidant effect of lactoferrin vs standard antioxidant drug (Acetyl cysteine) indicated by Anti-oxidant marker (TAC) 3- A comparison between the anti-inflammatory effect of lactoferrin vs standard anti-inflammatory, and immunomodulatory drug (dexamethasone) as indicated by the inflammatory marker (TNF- α)

3.5 Statistical analysis and sample size

Statistical analysis:

Per-protocol strategy will be used in this study. Categorical variables will be presented as proportion and percent. Continuous variables will be presented as mean (standard deviation) if normally distributed or as a median (IQR) or (25th-75th percentile) for non-normally distributed data Mann-Whitney test, t-test or Chi-square test will be used to compare baseline characteristics and outcomes between the two groups. In comparison between the two groups, Chi-square test will be used to compare proportions for non-parametric data (nominal or categorical). Mann-Whitney test will be used to compare medians for non- normally distributed continuous parametric data. While t-test will be used only to compare means in case normally distributed continuous parametric. So, distributions of continuous data will be tested in order to know the correct test to be used in comparison of parametric data between the two groups. ANOVA test will be used in case of comparison between more than 2 groups (as in case of comparison of antioxidant therapies).

Investigators will report the 95% confidence interval and the P-value for our statistical tests with level of statistical significance will be p-value < 0.05.

Regression analysis will be performed, if there is a statistically significant differences between the baseline characteristics including age, gender, No. of comorbidities (DM, hypertension (HTN), ischemic heart disease (IHD), atrial fibrillation (AF), COPD) in order to exclude the effect of these confounding variables on the study outcomes Investigators will compare the 28-day all-cause mortality rate, incidence of hypersensitivity reactions, and need for invasive mechanical ventilation (IMV) using the Chi-square test. while t-test will be used to compare the day of death, duration of need for oxygen therapy and IMV, and duration of ICU stay, and all parameter measured in the study if they will be normally distributed, but if they will be non-normally distributed, Mann-Whitney test will be used instead.

. Statistical analysis will be achieved with SPSS software, version 26.

Sample size:

The power of trial will depend on the primary outcome (28-day mortality). The proportion of ICU Population to all hospital population is about 25% A total sample sizes of 634 patients would achieve at least 80 % (0.8) power to detect a risk difference of 0.2 (20%) in the 28-day all-cause mortality (primary outcome) between alternative hypothesis and the null hypothesis (proportions of two groups are 0.5) with a significance level (α) of 0.05 and 95% confidence level proportion in Clincalc.com calculator [62]. To compensate for the estimated loss-to-follow-up and increase the study power more than 80%, Investigators will increase the sample size in both groups to be 660 patients (330 in each study group).

The mortality data will be estimated from the average mortality in January, February, and March 2025 at the Mansoura University Hospital ICU departments among all hospitalized patients. Mortality rate is found to be about 720 cases in these 3 months (240 cases / month) in ICU patients receiving the standard of care. The online system has been used to obtain mortality rate in these three months [32-39]. The hypothesis is that LF will decrease mortality by 20% so mortality rate will be decreased from 240 to 192 per month.

4. Data Quality and Safety

Investigators will collect the data from hospital system directly into an excel sheet, Patient confidentiality will be kept before, during and after the study. Patients who will be discharged before 28 days of hospital stay, will be communicated at day 28 in order to know mortality at day 28.

5. Publishing the study results and funding

Due to size limitations in publishing the research as one paper in a journal. Investigators aim to divide this research into five papers and publish these papers in peer-reviewed journals (5 stage publications).

Funding There is no funding source for this study

Conflict of interest The investigators declare no relevant conflict of interest

6. Ethical Considerations

Ethical approval will be taken from

1. Institutional research board (IRB), faculty of medicine, Mansoura University,
2. Research ethics committee, faculty of pharmacy, Tanta University,

   * Benefits of the intervention to the patients outweigh expected risks. Informed consents will be obtained from all participants in this research. Privacy of participants and the confidentiality of data will be maintained. Any unexpected risks that appeared during the research will be cleared to participants, the IRB, and ethical committees on time. All study procedures will obey the standard of the Declaration of Helsinki (1964) principles

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for patients to participate in this research include adult (age ≥ 18 years) patients admitted to ICU for any reason or disease.

Exclusion Criteria:

* inability to give informed consent by patients or their relative,
* history of hypersensitivity to milk products,
* history of lactoferrin use in the past 6 months,
* patients with lactose intolerance,
* patients with no enteral access to administer LF either orally or by Ryle tube,
* patients who are expected to die within 48 hours, and
* patients with poor oral absorption as in case of shock and resected bowel.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2027-12-29 (Estimated); Study Completion 2027-12-29 (Estimated)

PRIMARY OUTCOMES:
28-days mortality rate | 28 days
  Dead or alive
Number of Participants With any allergic or hypersensitivity reactions | up to 60 days
  incidence of any allergic or hypersensitivity reactions

SECONDARY OUTCOMES:
Day of death | up to 60 days
  Death day
Incidence of need for Invasive Mechanical Ventilation | up to 60 days
  yes or no
Oxygen Support Duration | up to 60 days
  Duration of need for Oxygen Support
Duration of ICU stay | up to 60 days
  ICU stay duration
White blood cells (WBCs) counts on day 3 | day 3
  Leukocytes count on day 3
White blood cells (WBCs) counts on day 7 | day 7
  Leukocytes count on day 7
White blood cells (WBCs) counts on day 14 | day 14
  Leukocytes count on day 14
White blood cells (WBCs) counts on day 28 | day 28
  Leukocytes count on day 28
Neutrophils counts on day 3 | day 3
  Neutrophils counts on day 3
Neutrophils counts on day 7 | day 7
  Neutrophils counts on day 7
Neutrophils counts on day 14 | day 14
  Neutrophils counts on day 14
Neutrophils counts on day 28 | day 28
  Neutrophils counts on day 28
Hemoglobin concentration on day 3 | day 3
  Hemoglobin concentration on day 3
Hemoglobin concentration on day 7 | day 7
  Hemoglobin concentration on day 7
Hemoglobin concentration on day 14 | day 14
  Hemoglobin concentration on day 14
Hemoglobin concentration on day 28 | day 28
  Hemoglobin concentration on day 28
Hematocrit concentration on day 3 | day 3
  Hematocrit concentration on day 3
Hematocrit concentration on day 7 | day 7
  Hematocrit concentration on day 7
Hematocrit concentration on day 14 | day 14
  Hematocrit concentration on day 14
Hematocrit concentration on day 28 | day 28
  Hematocrit concentration on day 28
Platelets counts on day 3 | day 3
  Platelets counts on day 3
Platelets counts on day 7 | day 7
  Platelets counts on day 7
Platelets counts on day 14 | day 14
  Platelets counts on day 14
Platelets counts on day 28 | day 28
  Platelets counts on day 28
Sequential Organ Function Assessment (SOFA) Score on day 3 | day 3
  minimum 0 to maximum 24, higher scores mean worse outcomes
Sequential Organ Function Assessment (SOFA) Score on day 7 | day 7
  minimum 0 to maximum 24, higher scores mean worse outcomes
Sequential Organ Function Assessment (SOFA) Score on day 14 | day 14
  minimum 0 to maximum 24, higher scores mean worse outcomes
Sequential Organ Function Assessment (SOFA) Score on day 28 | day 28
  minimum 0 to maximum 24, higher scores mean worse outcomes
Aspartate Aminotransferase (AST) concentration on day 3 | day 3
  Aspartate Aminotransferase (AST) concentration on day 3
Aspartate Aminotransferase (AST) concentration on day 7 | day 7
  Aspartate Aminotransferase (AST) concentration on day 7
Aspartate Aminotransferase (AST) concentration on day 14 | day 14
  Aspartate Aminotransferase (AST) concentration on day 14
Aspartate Aminotransferase (AST) concentration on day 28 | day 28
  Aspartate Aminotransferase (AST) concentration on day 28
Alanine Aminotransferase (ALT) concentration on day 3 | day 3
  Alanine Aminotransferase (ALT) concentration on day 3
Alanine Aminotransferase (ALT) concentration on day 7 | day 7
  Alanine Aminotransferase (ALT) concentration on day 7
Alanine Aminotransferase (ALT) concentration on day 14 | day 14
  Alanine Aminotransferase (ALT) concentration on day 14
Alanine Aminotransferase (ALT) concentration on day 28 | day 28
  Alanine Aminotransferase (ALT) concentration on day 28
Albumin concentration on day 3 | day 3
  Albumin concentration on day 3
Albumin concentration on day 7 | day 7
  Albumin concentration on day 7
Albumin concentration on day 14 | day 14
  Albumin concentration on day 14
Albumin concentration on day 28 | day 28
  Albumin concentration on day 28
Bilirubin concentration on day 3 | day 3
  Bilirubin concentration on day 3
Bilirubin concentration on day 7 | day 7
  Bilirubin concentration on day 7
Bilirubin concentration on day 14 | day 14
  Bilirubin concentration on day 14
Bilirubin concentration on day 28 | day 28
  Bilirubin concentration on day 28
Serum Creatinine (S.Cr) concentration on day 3 | day 3
  Serum Creatinine (S.Cr) concentration on day 3
Serum Creatinine (S.Cr) concentration on day 7 | day 7
  Serum Creatinine (S.Cr) concentration on day 7
Serum Creatinine (S.Cr) concentration on day 14 | day 14
  Serum Creatinine (S.Cr) concentration on day 14
Serum Creatinine (S.Cr) concentration on day 28 | day 28
  Serum Creatinine (S.Cr) concentration on day 28
Creatinine clearance (Cr.Cl) rate on day 3 | day 3
  Creatinine clearance (Cr.Cl) rate on day 3
Creatinine clearance (Cr.Cl) rate on day 7 | day 7
  Creatinine clearance (Cr.Cl) rate on day 7
Creatinine clearance (Cr.Cl) rate on day 14 | day 3
  Creatinine clearance (Cr.Cl) rate on day 14
Creatinine clearance (Cr.Cl) rate on day 28 | day 28
  Creatinine clearance (Cr.Cl) rate on day 28
Duration of hospitalization | up to 60 days
  Duration of hospitalization
Antioxidant marker at day 14 | Bi-weekly
  Total Antioxidant Capacity (TAC)
Antioxidant marker at day 28 | Bi-weekly
  Total Antioxidant Capacity (TAC)
Inflammatory marker at day 14 | Bi-weekly
  TNF-alpha
Inflammatory marker at day 28 | Bi-weekly
  TNF- alpha

OTHER OUTCOMES:
Glasgow Coma Score (GCS) on day 3 | day 3
  minimum 0 to maximum 15, higher scores mean better outcomes
Glasgow Coma Score (GCS) on day 7 | day 7
  minimum 0 to maximum 15, higher scores mean better outcomes
Glasgow Coma Score (GCS) on day 14 | day 14
  minimum 0 to maximum 15, higher scores mean better outcomes
Glasgow Coma Score (GCS) on day 28 | day 28
  minimum 0 to maximum 15, higher scores mean better outcomes
Arterial Oxygen Pressure / Fraction Inspired of Oxygen (PaO2/FiO2) on day 3 | day 3
  Arterial Oxygen Pressure / Fraction Inspired of Oxygen (PaO2/FiO2) on day 3
Arterial Oxygen Pressure / Fraction Inspired of Oxygen (PaO2/FiO2) on day 7 | day 7
  Arterial Oxygen Pressure / Fraction Inspired of Oxygen (PaO2/FiO2) on day 7
Arterial Oxygen Pressure / Fraction Inspired of Oxygen (PaO2/FiO2) on day 14 | day 14
  Arterial Oxygen Pressure / Fraction Inspired of Oxygen (PaO2/FiO2) on day 14
Arterial Oxygen Pressure / Fraction Inspired of Oxygen (PaO2/FiO2) on day 28 | day 28
  Arterial Oxygen Pressure / Fraction Inspired of Oxygen (PaO2/FiO2) on day 28
Oxygen saturation on day 3 | day 3
  Oxygen saturation at day 3
Oxygen saturation on day 7 | day 7
  Oxygen saturation at day 7
Oxygen saturation on day 14 | day 14
  Oxygen saturation at day 14
Oxygen saturation on day 28 | day 28
  Oxygen saturation at day 28

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H Hassan, Pharmacist, Principal Investigator — Mansoura University Hospital
Locations (1):
- Mansoura University hospital, Al Mansurah, El-dakhlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After the end and publication of the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the end and publication of the study
Access Criteria: all will be accessible
URL: https://drive.google.com/drive/folders/1CBAPVtAVYsi2x1iLQdWl48b9OowGSxw9

REFERENCES:
- [Background] Artym J, Kocieba M, Zaczynska E, Adamik B, Kubler A, Zimecki M, Kruzel M. Immunomodulatory properties of human recombinant lactoferrin in mice: Implications for therapeutic use in humans. Adv Clin Exp Med. 2018 Mar;27(3):391-399. doi: 10.17219/acem/68440. PMID 29533543
- [Background] Hegazy, S.K., Hassan, A.H. The effect of combination treatment with casirivimab and imdevimab versus standard antiviral therapy on clinical outcomes in hospitalized COVID-19 patients. Discov Med 1, 71 (2024). https://doi.org/10.1007/s44337-024-00045-3
- [Background] Baker HM, Baker EN. A structural perspective on lactoferrin function. Biochem Cell Biol. 2012 Jun;90(3):320-8. doi: 10.1139/o11-071. Epub 2012 Jan 31. PMID 22292559
- [Background] Legrand D, Pierce A, Elass E, Carpentier M, Mariller C, Mazurier J. Lactoferrin structure and functions. Adv Exp Med Biol. 2008;606:163-94. doi: 10.1007/978-0-387-74087-4_6. PMID 18183929
- [Background] Siqueiros-Cendon T, Arevalo-Gallegos S, Iglesias-Figueroa BF, Garcia-Montoya IA, Salazar-Martinez J, Rascon-Cruz Q. Immunomodulatory effects of lactoferrin. Acta Pharmacol Sin. 2014 May;35(5):557-66. doi: 10.1038/aps.2013.200. PMID 24786230
- [Background] Bukowska-Osko I, Popiel M, Kowalczyk P. The Immunological Role of the Placenta in SARS-CoV-2 Infection-Viral Transmission, Immune Regulation, and Lactoferrin Activity. Int J Mol Sci. 2021 May 28;22(11):5799. doi: 10.3390/ijms22115799. PMID 34071527
- [Background] Kowalczyk P, Kaczynska K, Kleczkowska P, Bukowska-Osko I, Kramkowski K, Sulejczak D. The Lactoferrin Phenomenon-A Miracle Molecule. Molecules. 2022 May 4;27(9):2941. doi: 10.3390/molecules27092941. PMID 35566292
- [Background] Poljsak B, Suput D, Milisav I. Achieving the balance between ROS and antioxidants: when to use the synthetic antioxidants. Oxid Med Cell Longev. 2013;2013:956792. doi: 10.1155/2013/956792. Epub 2013 Apr 29. PMID 23738047
- [Background] Kowalczyk P, Sulejczak D, Kleczkowska P, Bukowska-Osko I, Kucia M, Popiel M, Wietrak E, Kramkowski K, Wrzosek K, Kaczynska K. Mitochondrial Oxidative Stress-A Causative Factor and Therapeutic Target in Many Diseases. Int J Mol Sci. 2021 Dec 13;22(24):13384. doi: 10.3390/ijms222413384. PMID 34948180
- [Background] Parekattil S.J., Esteves S.C., Agarwal A. Male Infertility. Springer; Berlin/Heidelberg, Germany: 2020. Harmful Effects of Antioxidant Therapy
- [Background] Abdelhamid M, Jung CG, Zhou C, Abdullah M, Nakano M, Wakabayashi H, Abe F, Michikawa M. Dietary Lactoferrin Supplementation Prevents Memory Impairment and Reduces Amyloid-beta Generation in J20 Mice. J Alzheimers Dis. 2020;74(1):245-259. doi: 10.3233/JAD-191181. PMID 31985470
- [Background] Shi P, Fan F, Chen H, Xu Z, Cheng S, Lu W, Du M. A bovine lactoferrin-derived peptide induced osteogenesis via regulation of osteoblast proliferation and differentiation. J Dairy Sci. 2020 May;103(5):3950-3960. doi: 10.3168/jds.2019-17425. Epub 2020 Mar 18. PMID 32197844
- [Background] Moreno-Navarrete JM, Ortega FJ, Bassols J, Ricart W, Fernandez-Real JM. Decreased circulating lactoferrin in insulin resistance and altered glucose tolerance as a possible marker of neutrophil dysfunction in type 2 diabetes. J Clin Endocrinol Metab. 2009 Oct;94(10):4036-44. doi: 10.1210/jc.2009-0215. Epub 2009 Jul 7. PMID 19584176
- [Background] Kaczmarek N, Jamka M, Walkowiak J. [An association of selected polymorphisms of the lactoferrin gene and genes for lactoferrin receptors in the prevalence of metabolic disorders in obese subjects]. Pol Merkur Lekarski. 2020 Apr 22;48(284):120-123. Polish. PMID 32352945
- [Background] Ikeda Y, Tajima S, Izawa-Ishizawa Y, Kihira Y, Ishizawa K, Yoshida S, Aihara K, Tsuchiya K, Tamaki T. Bovine milk-derived lactoferrin exerts proangiogenic effects in an Src-Akt-eNOS-dependent manner in response to ischemia. J Cardiovasc Pharmacol. 2013 May;61(5):423-9. doi: 10.1097/FJC.0b013e318287d526. PMID 23364610
- [Background] Jenssen H, Hancock RE. Antimicrobial properties of lactoferrin. Biochimie. 2009 Jan;91(1):19-29. doi: 10.1016/j.biochi.2008.05.015. Epub 2008 Jun 5. PMID 18573312
- [Background] Artym J, Zimecki M. Milk-derived proteins and peptides in clinical trials. Postepy Hig Med Dosw (Online). 2013 Aug 6;67:800-16. doi: 10.5604/17322693.1061635. PMID 24018446
- [Background] Tolone S, Pellino V, Vitaliti G, Lanzafame A, Tolone C. Evaluation of Helicobacter Pylori eradication in pediatric patients by triple therapy plus lactoferrin and probiotics compared to triple therapy alone. Ital J Pediatr. 2012 Oct 31;38:63. doi: 10.1186/1824-7288-38-63. PMID 23114016
- [Background] Wu J, Chen J, Wu W, Shi J, Zhong Y, van Tol EA, Tang Q, Cai W. Enteral supplementation of bovine lactoferrin improves gut barrier function in rats after massive bowel resection. Br J Nutr. 2014 Aug 28;112(4):486-92. doi: 10.1017/S000711451400107X. Epub 2014 May 15. PMID 24830343
- [Background] Sherman MP, Sherman J, Arcinue R, Niklas V. Randomized Control Trial of Human Recombinant Lactoferrin: A Substudy Reveals Effects on the Fecal Microbiome of Very Low Birth Weight Infants. J Pediatr. 2016 Jun;173 Suppl:S37-42. doi: 10.1016/j.jpeds.2016.02.074. PMID 27234409
- [Background] Berlutti F, Pantanella F, Natalizi T, Frioni A, Paesano R, Polimeni A, Valenti P. Antiviral properties of lactoferrin--a natural immunity molecule. Molecules. 2011 Aug 16;16(8):6992-7018. doi: 10.3390/molecules16086992. PMID 21847071
- [Background] Miotto M, Di Rienzo L, Bo L, Boffi A, Ruocco G, Milanetti E. Molecular Mechanisms Behind Anti SARS-CoV-2 Action of Lactoferrin. Front Mol Biosci. 2021 Feb 15;8:607443. doi: 10.3389/fmolb.2021.607443. eCollection 2021. PMID 33659275
- [Background] Manzoni P, Stolfi I, Messner H, Cattani S, Laforgia N, Romeo MG, Bollani L, Rinaldi M, Gallo E, Quercia M, Maule M, Mostert M, Decembrino L, Magaldi R, Mosca F, Vagnarelli F, Memo L, Betta PM, Stronati M, Farina D; Italian Task Force for the Study and Prevention of Neonatal Fungal Infections-the Italian Society of Neonatology. Bovine lactoferrin prevents invasive fungal infections in very low birth weight infants: a randomized controlled trial. Pediatrics. 2012 Jan;129(1):116-23. doi: 10.1542/peds.2011-0279. Epub 2011 Dec 19. PMID 22184648
- [Background] León-Sicairos N., Ordaz-Pichardo C., Carrero J.C., de la Garza M. Natural Remedies in the Fight Against Parasites. Intechopen; London, UK: 2017. Lactoferrin in the Battle against Intestinal Parasites: A Review.
- [Background] Yamauchi K, Wakabayashi H, Shin K, Takase M. Bovine lactoferrin: benefits and mechanism of action against infections. Biochem Cell Biol. 2006 Jun;84(3):291-6. doi: 10.1139/o06-054. PMID 16936799
- [Background] Alexander DB, Iigo M, Abdelgied M, Ozeki K, Tanida S, Joh T, Takahashi S, Tsuda H. Bovine lactoferrin and Crohn's disease: a case study. Biochem Cell Biol. 2017 Feb;95(1):133-141. doi: 10.1139/bcb-2016-0107. Epub 2016 Nov 30. PMID 28165294
- [Background] He S, McEuen AR, Blewett SA, Li P, Buckley MG, Leufkens P, Walls AF. The inhibition of mast cell activation by neutrophil lactoferrin: uptake by mast cells and interaction with tryptase, chymase and cathepsin G. Biochem Pharmacol. 2003 Mar 15;65(6):1007-15. doi: 10.1016/s0006-2952(02)01651-9. PMID 12623133
- [Background] Wakabayashi H, Yamauchi K, Abe F. Quality control of commercial bovine lactoferrin. Biometals. 2018 Jun;31(3):313-319. doi: 10.1007/s10534-018-0098-2. Epub 2018 Apr 4. PMID 29619653
- [Background] Nappi C, Tommaselli GA, Morra I, Massaro M, Formisano C, Di Carlo C. Efficacy and tolerability of oral bovine lactoferrin compared to ferrous sulfate in pregnant women with iron deficiency anemia: a prospective controlled randomized study. Acta Obstet Gynecol Scand. 2009;88(9):1031-5. doi: 10.1080/00016340903117994. PMID 19639462
- [Background] Chang R, Ng TB, Sun WZ. Lactoferrin as potential preventative and adjunct treatment for COVID-19. Int J Antimicrob Agents. 2020 Sep;56(3):106118. doi: 10.1016/j.ijantimicag.2020.106118. Epub 2020 Jul 30. PMID 32738305
- [Background] Vincent JL, de Mendonca A, Cantraine F, Moreno R, Takala J, Suter PM, Sprung CL, Colardyn F, Blecher S. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998 Nov;26(11):1793-800. doi: 10.1097/00003246-199811000-00016. PMID 9824069
- [Background] Eltahan NH, Elsawy NH, Abdelaaty KM, Elhamaky AS, Hassan AH, Emara MM. Atorvastatin for reduction of 28-day mortality in severe and critical COVID-19 patients: a randomized controlled trial. Respir Res. 2024 Feb 22;25(1):97. doi: 10.1186/s12931-024-02732-2. PMID 38389078
- [Background] Hegazy SK, Tharwat S, Hassan AH. Clinical study to compare the efficacy and safety of casirivimab & imdevimab, remdesivir, and favipravir in hospitalized COVID-19 patients. J Clin Virol Plus. 2023 Jun;3(2):100151. doi: 10.1016/j.jcvp.2023.100151. Epub 2023 May 10. PMID 37220480
- [Background] Hegazy SK, Tharwat S, Hassan AH. Study to compare the effect of casirivimab and imdevimab, remdesivir, and favipiravir on progression and multi-organ function of hospitalized COVID-19 patients. Open Med (Wars). 2023 Aug 9;18(1):20230768. doi: 10.1515/med-2023-0768. eCollection 2023. PMID 37588660
- [Background] Hegazy SK, Tharwat S, Hassan AH. Comparing the efficacy of regen-cov, remdesivir, and favipiravir in reducing invasive mechanical ventilation need in hospitalized COVID-19 patients. World J Clin Cases. 2023 Sep 16;11(26):6105-6121. doi: 10.12998/wjcc.v11.i26.6105. PMID 37731581
- [Background] Hegazy SK, Hassan AH. Comparing the Efficacy of Remdesivir, Favipiravir, and Casirivimab and Imdevimab on Duration of Hospitalization and ICU Stay of Hospitalized COVID-19 Patients. Life Science Research Communications; 2024; 1(1),21-30. Available at: https://doi.org/10.5530/lsrc.1.1.7
- [Background] Hassan AH, Hegazy SK, Radwan ST. Clinical Study to Evaluate the Possible Efficacy and Safety of Antibodies Combination (casirivimab and imdevimab) versus standard antiviral therapy as antiviral agent against Corona virus 2 infection in hospitalized COVID-19 patients. medRxiv. 2022. (preprint). Available from: doi: 10.1101/2022.08.20.22279020
- [Background] Hassan AH, Hegazy SK, Radwan ST. Clinical Study to Evaluate the Possible Efficacy and Safety of Antibodies Combination (casirivimab and imdevimab) versus standard antiviral therapy as antiviral agent against Corona virus 2 infection in hospitalized COVID-19 patients. Research Square; 2023. Available from: doi: 10.21203/rs.3.rs-1991618/v2.
- See also: Study data — https://drive.google.com/drive/folders/1CBAPVtAVYsi2x1iLQdWl48b9OowGSxw9
- Available data/document: Individual Participant Data Set — https://drive.google.com/drive/folders/1CBAPVtAVYsi2x1iLQdWl48b9OowGSxw9